CLINICAL TRIAL: NCT05507606
Title: Phase I Study of Osimertinib+Bevacizumab+Carboplatin and Pemetrexed for Untreated Patients With EGFR Mutation Advanced Non-squamous Non-Small Cell Lung Cancer With Concomitant Mutations.
Brief Title: Study of Osimertinib+Bevacizumab+Chemotherapy for EGFR+ Advanced Non-Small Cell Lung Cancer With Concurrent Mutations
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20210961
Record Dates: First submitted 2022-08-16; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Non Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; Angiogenesis Inhibitors; Carboplatin; Drug Therapy; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osimertinib+Bevacizumab+Carboplatin and Pemetrexed (Experimental): Bevacizumab, 7.5mg/kg, d1; Pemetrexed, 500mg/m2, d1; Carboplatin AUC5, d1; Osimertinib 80mg/d , d1-21; Q3W/cycle induction therapy for 4 cycle. Then Carboplatin was stopped after 4 cycles, and Osimertinib combined with Bevacizumab and Pemetrexed were given for maintenance treatment every 3 weeks for 2 years. After that, the maintenance treatment of Osimertinib was continued.
  Interventions: Drug: Osimertinib; Drug: Bevacizumab Biosimilar IBI305; Drug: Carboplatin; Drug: Pemetrexed

INTERVENTIONS:
Drug: Osimertinib — osimertinib 80mg/d
  Other Names: EGFR-TKI
Drug: Bevacizumab Biosimilar IBI305 — Bevacizumab, 7.5mg/kg d1; was discontinued after 2 years
  Other Names: Anti-angiogenesis
Drug: Carboplatin — Carboplatin AUC5, d1; was stopped after 4 cycles
  Other Names: Chemotherapy
Drug: Pemetrexed — Pemetrexed, 500mg/m2, d1;Q3W/cycle; was discontinued after 2 years
  Other Names: Chemotherapy

SUMMARY:
This is a single-center, open-label, phase I clinical trial aimed to evaluate the efficacy and safety of Osimertinib+Bevacizumab+Carboplatin and Pemetrexed for Untreated Patients With EGFR Mutation Advanced Non-squamous Non-Small Cell Lung Cancer With Concomitant Mutations.

DETAILED DESCRIPTION:
Patients received Bevacizumab, 7.5mg/kg d1, Pemetrexed, 500mg/m2, d1 and Carboplatin AUC5, d1; osimertinib 80mg/d , d1-21, Q3W/cycle; induction therapy for 4 cycle, then Carboplatin was stopped after 4 cycles, and osimertinib combined with bevacizumab and pemetrexed were given for maintenance treatment every 3 weeks; Bevacizumab and pemetrexed were discontinued for 2 years; After that, the maintenance treatment of osimertinib was continued

ELIGIBILITY:
Inclusion Criteria:

Subjects who must meet all the following criteria should be selected:

1. Agree to participate in this trial and sign written informed consent form.
2. Male or female, age between 18 and 70 years.
3. Expected survival time ≥ 3 months and able to be followed-up.
4. Stage IIIB/IIIC/IV non-squamous NSCLC patients without previous systemic therapy (according to AJCC8th) or patients with stage IIIB/IIIC/IV non-squamous NSCLC who have relapsed after surgery (if adjuvant therapy was administered, more than 6 months of drug discontinuation is required).
5. The tumor harbors epidermal growth factor receptor (EGFR) mutations(include 19del, L858R, T790M, G719X, L861Q, S768I, 20 A763-Y764ins), and at least concurrent with TP53
6. Patients can not receive concurrent chemoradiothrapy after multidisciplinary consultation and discussion.
7. At least one measurable tumor indicator along with a lesion with a maximum diameter of ≥ 1 cm (diagnosed by imaging, e.g., CT, MRI, ECT).
8. ECOG PS 0-1 within 7 days before enrollment.
9. Within 14 days prior to the start of treatment, laboratory results of routine blood, liver and kidney function and hormone levels meet the following criteria: white blood cell(WBC) ≥3.5× 109/L, platelets (PLT) ≥ 80 × 109/L, neutrophils (ANC) ≥ 1.5 × 109/L, hemoglobin (HGB) ≥ 80 g/L, aspartate aminotransferase (AST) ≤ 2.5 × upper limit of normal (ULN) (≤ 5 × ULN for liver metastases), alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for liver metastases), total bilirubin (TIBC) ≤ 1.5 × ULN, and alanine aminotransferase (ALT) ≤ 1.5 × ULN. × ULN), alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 × ULN for liver metastases), total bilirubin (TIBC) ≤ 1.5 × ULN, serum creatinine (CR) ≤ 1.25 × ULN; cortisol and thyroid function are in the normal range.
10. Toxic effects of prior chemotherapy have resolved to grade 1 or less (except alopecia). Subjects must have recovered from toxicity or complications of these interventions if they have received major surgical treatment or > 30Gy of radiation therapy, i.e., they are still eligible for enrollment after 6 months.

Exclusion Criteria:

Subjects who meet any of the following criteria could not participate in this study:

1. non-squamous NSCLC just harbors EGFR mutations
2. Prior treatment with first,second and 3rd EGFR-TKI.
3. Received bevacizumab and/or pemetrexed within 6 months prior to the first dose of study drug.
4. Prior treatment with PD-1/PD-L1 antibodies within 3 months prior to the first dose of study drug.
5. Received anti-tumor monoclonal antibody (mAb), chemotherapy, targeted small molecule therapy, or major surgical procedure within 1 month prior to the first use of study drug; received chest radiation therapy greater than 30 Gy within 6 months prior to the first use of study drug; received chest radiation therapy at 30 Gy or less within 1 month prior to the first use of study drug.
6. Participating or have participated in investigational drug therapy within 4 weeks prior to the first dose of the trial.
7. Other malignant tumors with disease progression or requiring aggressive treatment within 5 years of enrollment. Exceptions included early-stage tumors (carcinoma in situ or stage I tumors) that received radical treatment, basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, or carcinoma in situ of the breast that received potentially radical treatment.
8. Having congenital or acquired immune deficiency (e.g., HIV-infected patients), active hepatitis B (HBV-DNA ≥10^3 copies/ml), or hepatitis C (positive for hepatitis C antibodies and HCV-RNA above the lower limit of detection for the assay).
9. Patients who have received live vaccine within 4 weeks prior to the first administration of study drug are permitted to receive inactivated viral.
10. Patients with known active central nervous system (CNS) metastases and/or cancerous meningitis. Subjects who have had treatment for brain metastases may also participate in this study provided that the subject is stable (no evidence of progression for at least 4 weeks and all neurological symptoms have returned to baseline levels as determined by MRI prior to the first dose), has no evidence of new or expanding brain metastases, and has not used hormone therapy for at least 3 days prior to study dosing.
11. Bleeding tendency, high bleeding risk, or coagulopathy with a history of thrombotic disease within 6 months and/or hemoptysis within 3 months; being treated with full doses of oral and/or parenteral anticoagulants and thrombolytics (prophylactic anticoagulation is allowed); having used aspirin or other non-steroidal anti-inflammatory drugs that inhibit platelet function within 10 days; and CT/MRI imaging showing tumor encapsulation or invasion of the lumen of large blood vessels.
12. Poorly controlled hypertension (systolic >150 mmHg and/or diastolic >100 mmHg) and patients with prior hypertensive crisis and hypertensive encephalopathy; severe cerebrovascular disease.
13. Non-healing wounds, peptic ulcers in active phase, tracheo-esophageal fistulas, gastrointestinal perforations and intra-abdominal abscesses within 6 months.
14. Have an active infection that requires systemic treatment via Intravenous injection.
15. Have mental illness or other condition, such as uncontrolled heart or lung disease, diabetes mellitus, etc., that prevents cooperation with study treatment and monitoring requirements.
16. Known allergy to any of the components of the study drug.
17. Patients who are regular users of any drug (including "recreational" use) or have recent history (within 1 year) of substance abuse (including alcohol) when signing the informed consent form.
18. Pregnancy or breast feeding.
19. Poor compliance and inability to cooperate with the clinical study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 2 years
  ORR was calculated by the percentage of patients with a confirmed complete (CR) or partial response (PR).

SECONDARY OUTCOMES:
OS | 3 years
  Time from the first use of the study drug to the death of the subject
PFS | 2 years
  Progression-free survival is defined as the time from the start of treatment to the first documentation of disease progression or death from any cause, whichever occurs first according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol